CLINICAL TRIAL: NCT02567500
Title: Identification of Cognitive and Emotional Factors in Relation to Auditory Hallucinations in Non-psychotic Children
Brief Title: The Physalis Child : Identification of Cognitive and Emotional Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-HPNCL-02
Record Dates: First submitted 2015-07-24; First posted 2015-10-05 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Auditory Hallucinations
Keywords: emotional; auditory hallucinations; non-psychotic children
MeSH Terms: conditions — Hallucinations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with auditory hallucination (Experimental): Patients with auditory hallucination:
  Evaluation at time 0 and 6 month after of:
  * The social cognitive marker (NeuroPsychologic assessment (NEPSY) II) : theory of mind and affect recognition
  * The emotional marker:
    * Differential Emotion Scale IV (DES IV): emotional individual stability
    * Revised Beliefs About Voices Questionnaire (BAVQ-R): a self report measure of patients' beliefs, emotional and behavior about auditory hallucination.
  * Evaluation of auditory hallucinations persistence with a self report scale using in recruiting criteria.
  * Evaluation of diagnosis with Diagnostic and Statistical Manual of Mental Disorders (DSM) -IV criteria:
    * Mini International Neuropsychiatric Interview (MINI) -Kids
    * "Psychosis" section of Kiddie-SADS
  Interventions: Behavioral: Patients with auditory hallucination
- Patients without auditory hallucination (Placebo Comparator): Patients without auditory hallucination:
  Evaluation at time 0 and 6 month after of:
  * The social cognitive marker (NEPSY II) : theory of mind and affect recognition
  * The emotional marker:
    * Differential emotion scale IV (DES IV): emotional individual stability
    * Revised Beliefs About Voices Questionnaire (BAVQ-R): a self report measure of patients' beliefs, emotional and behavior about auditory hallucination.
  * Evaluation of auditory hallucinations persistence with a self report scale using in recruiting criteria.
  * Evaluation of diagnosis with Diagnostic and Statistical Manual of Mental Disorders (DSM) -IV criteria:
    * Mini International Neuropsychiatric Interview (MINI) -Kids
    * "Psychosis" section of Kiddie-SADS (Schedule for Affective Disorders and Schizophrenia )
  Interventions: Behavioral: Patients without auditory hallucination

INTERVENTIONS:
Behavioral: Patients with auditory hallucination — Patients with auditory hallucination (20 for each arm):
  Evaluation at time 0 and 6 month after of:
  * The social cognitive marker (NEPSY II) : theory of mind and affect recognition
  * The emotional marker:
    * Differential emotion scale IV (DES IV): emotional individual stability
    * Revised Beliefs About Voices Questionnaire (BAVQ-R): a self report measure of patients' beliefs, emotional and behavior about auditory hallucination.
  * Evaluation of auditory hallucinations persistence with a self report scale using in recruiting criteria.
  * Evaluation of diagnosis with DSM-IV criteria:
    * MINI-Kids
    * "Psychosis" section of Kiddie-SADS
  Arms: Patients with auditory hallucination
Behavioral: Patients without auditory hallucination — Patients without auditory hallucination (20 for each arm):
  Evaluation at time 0 and 6 month after of:
  * The social cognitive marker (NEPSY II) : theory of mind and affect recognition
  * The emotional marker:
    * Differential emotion scale IV (DES IV): emotional individual stability
    * Revised Beliefs About Voices Questionnaire (BAVQ-R): a self report measure of patients' beliefs, emotional and behavior about auditory hallucination.
  * Evaluation of auditory hallucinations persistence with a self report scale using in recruiting criteria.
  * Evaluation of diagnosis with DSM-IV criteria:
    * MINI-Kids
    * "Psychosis" section of Kiddie-SADS
  Arms: Patients without auditory hallucination

SUMMARY:
The aim of this study is to show presence of cognitive and emotional factors on the beginning and persistence of auditory hallucinations in non-psychotic children. Investigators will describe a significant link between this factors and hallucinations in a sample of non-psychotic children. The results of this sample will be comparing to another group of children of the same age, sex and diagnosis, but without hallucination. Finally, investigators will control the persistence of hallucination on the first group after a six month period.

DETAILED DESCRIPTION:
Background: Hallucinations are a common symptom in pediatric population without psychotic syndrome. Vulnerability, co morbidity and risk factor are already been described. Investigators will study the cognitive and emotional factors on the beginning and persistence of auditory hallucinations in non-psychotic children. The goal of the study is to find a social cognition our emotional impairment to explain auditory hallucinations without psychotic symptoms. Methods: Sample of out non-psychotic patients aged six to eighteen years old with auditory hallucinations were recruited with a self report scale created for this study. Mini International Neuropsychiatric Interview (MINI)-kids interview and "psychosis" section od Kiddie-SADS (Schedule for Affective Disorders and Schizophrenia for school age chidlren) were conducted to determine Diagnostic and Statistical Manual of Mental Disorders (DSM) IV diagnoses. All children patient were spend specifics social cognition (NeuroPsychologic assessment NEPSY II) and emotional (ifferential Emotions Scale (DES) IV, Beliefs About Voices Questionnaire Revised (BAVQ-R)) scales. Each child results will be compared to child result of the same age, sex and diagnosis but without hallucination that passed the same specifics scales. All of child will be control after a six month period to evaluate auditory hallucination persistence and diagnosis evolution. The total period of the study will be twelve month.

ELIGIBILITY:
Inclusion Criteria:

* Twenty participants included with auditory hallucination:

  * Boy or girl
  * French
  * Over six years old and under eighteen years old
  * DSM-IV diagnosis of mood disorder, anxiety, disruptive behavioral disorder, attention deficit hyperactivity disorder, without schizophrenia diagnosis, without mental retardation (Intelligence Quotient (IQ)>70),
  * Parental and child consent, affiliated to social security.
* Twenty participants included without auditory hallucination:

  * Boy or girl
  * French,
  * Over six years old and under eighteen years old
  * DSM-IV diagnosis of mood disorder, anxiety, disruptive behavioral disorder, attention deficit hyperactivity disorder, without schizophrenia diagnosis, without mental retardation (IQ>70)
  * Parental and child consent, affiliated to social security.

Exclusion Criteria:

* schizophrenia diagnosis,
* neurologic, genetic or neurosensory disorders

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Evolution of the score of theory of mind | Change from baseline 6 month later
  The social cognitive marker will be evaluate by NeuroPsychologic assessment NEPSY II for theory of mind

SECONDARY OUTCOMES:
Evolution of the score of auditory hallucinations persistence | Change from baseline 6 month later
  Evaluation of auditory hallucinations persistence with a self report scale using in recruiting criteria.
Evolution of the score of Mental Disorder | Change from baseline 6 month later
  Evaluation of diagnosis of Mental Disorder with Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV criteria using MINI-Kids (Mini International Neuropsychiatric Interview )
Evaluation of the score of Psychosis | Change from baseline 6 month later
  Evaluation of diagnosis of psychosis with DSM-IV (Diagnostic and Statistical Manual of Mental Disorders ) criteria using "Psychosis" section of Kiddie-SADS (Schedule for Affective Disorders and Schizophrenia for school age chidlren)
Evolution of the score of individual stability | Change from baseline 6 month later
  The evaluation of the the emotional marker will be performed with the Differential emotion scale IV (DES IV): emotional individual stability
Evolution of measure of recognition of the feelings | Change from baseline 6 month later
  The measure of recognition of the feelings will be performed by the score:
  The social cognitive marker (NEPSY II)
Evolution of auditory measure of patients' emotional | Change from baseline 6 month later
  The auditory measure will be performed by the score:
  The social cognitive marker (NEPSY II)
Evolution of Emotional real-life experience of the hallucination | Change from baseline 6 month later
  The Emotional real-life experience of the hallucination will be performed by the score:
  The Revised Beliefs About Voices Questionnaire (BAVQ-R)
Evolution of the score of affect recognition | Change from baseline 6 month later
  The social cognitive marker will be evaluate by NeuroPsychologic assessment NEPSY II for theory of affect recognition

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BONNARD-COUTON, MD, Principal Investigator — Fondation Lenval
Locations (1):
- Fondation Lenval, Nice, France

REFERENCES:
- [Derived] Dumas LE, Bonnard-Couton V, Golse B, Askenazy F. [Identifying cognitive and emotional markers in relation to auditory-verbal hallucinations in pediatric population: Physalis study]. Encephale. 2022 Oct;48(5):546-554. doi: 10.1016/j.encep.2021.06.010. Epub 2021 Oct 5. French. PMID 34625214